CLINICAL TRIAL: NCT01588782
Title: An Open-Label Drug-Drug Interaction Study to Assess the Effect of Ketoconazole on the Pharmacokinetics of Abiraterone (JNJ-589485) Following Administration of Abiraterone Acetate (JNJ-212082) Tablets in Healthy Male Subjects
Brief Title: A Study to Assess the Effect of Ketoconazole on the Pharmacokinetics of Abiraterone Following Administration of Abiraterone Acetate Tablets in Healthy Adult Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR100650; 212082PCR1002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2012-01-09; First posted 2012-05-01 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers; Pharmacology; Pharmacokinetics; Pharmacodynamics; Drug-drug interactions; CYP3A4; Abiraterone acetate; JNJ-589485; JNJ-212082; Ketoconazole
MeSH Terms: interventions — Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abiraterone acetate (Experimental): All individuals will receive study treatment in the same sequence. Period 1 (Days 1 to 4) consists of a single oral dose of 1000 mg abiraterone acetate tablets on Day 1 only. Period 2 (Days 11 to 17) consists of a daily oral dose of 400 mg ketoconazole tablets on Days 11 to 16 and administration of a single dose of 1000 mg abiraterone acetate on Day 14.
  Interventions: Drug: Period 1: Abiraterone; Drug: Period 2: Abiraterone/Ketoconazole

INTERVENTIONS:
Drug: Period 1: Abiraterone — 1000 mg abiraterone acetate tablet administered orally on Day 1
Drug: Period 2: Abiraterone/Ketoconazole — 400 mg ketoconazole tablets administered orally on Days 11 to 16
Drug: Period 2: Abiraterone/Ketoconazole — 1000 mg abiraterone acetate tablet administered orally on Day 14

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics, safety, and potential for drug-drug interactions when a strong inhibitor of CYP3A4 (ie, ketoconazole) is co-administered with abiraterone acetate in healthy adult men.

DETAILED DESCRIPTION:
This is a non-randomized (individuals will not be assigned by chance to study treatments), open-label (individuals will know the identity of study treatments), 2-period, sequential-design, drug-drug interaction study of abiraterone acetate and ketoconazole in approximately 20 healthy adult men. This study will consist of a screening period followed by an open-label treatment phase consisting of 2 treatment periods. Successive drug administration will be separated by a washout period of at least 10 days. All individuals will receive study treatment in the same sequence. Period 1 (Days 1 to 4) consists of a single oral dose of 1000 mg abiraterone acetate tablets on Day 1 only. Period 2 (Days 11 to 17) consists of a daily oral dose of 400 mg ketoconazole tablets on Days 11 to 16 and administration of a single dose of 1000 mg abiraterone acetate on Day 14. Serial pharmacokinetic (study of what the body does to a drug) samples will be collected at each treatment period as detailed in the protocol. Safety will be monitored continuously from the time of informed consent signing until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

- Body mass index (BMI) between 18 and 30 kg/m2, inclusive

Exclusion Criteria:

- History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Mean plasma concentrations of abiraterone | Up to Day 17
Mean plasma concentrations of ketoconazole | Up to Day 14
Maximum plasma concentrations of abiraterone | Up to Day 17
Time to reach the maximum plasma concentration of abiraterone | Up to Day 17
Area under the plasma concentration-time curve from time 0 to time to the last quantifiable concentration of abiraterone | Up to Day 17
Area under the plasma concentration-time curve from time 0 to infinite time of abiraterone | Up to Day 17
Elimination half-life associated with the terminal slope of the semilogarithmic drug concentration-time curve of abiraterone | Up to Day 17
First-order rate constant associated with the terminal portion of the curve of abiraterone | Up to Day 17
Time to last quantifiable plasma concentration of abiraterone | Up to Day 17
Percentage of area under the plasma concentration-time curve from time 0 to infinite time obtained by extrapolation of abiraterone | Up to Day 17

SECONDARY OUTCOMES:
The number of participants affected by an adverse event | Up to end of study or early withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium